CLINICAL TRIAL: NCT01947244
Title: Illinois Maternal, Infant, and Early Childhood Home Visiting (MIECHV): Doula Randomized Controlled Trial
Brief Title: Doula Home Visiting Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); Illinois Department of Human Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D89MC23146
Record Dates: First submitted 2013-09-13; First posted 2013-09-20 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Breast Feeding; Parenting; Child Development; Depression, Postpartum
Keywords: Doulas; Parenting; Breast Feeding; Pregnancy in Adolescence; Child Development
MeSH Terms: conditions — Breast Feeding; Depression, Postpartum | interventions — Case Management

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Doula Home Visiting (Experimental): Participants assigned to the intervention group receive prenatal and short-term postpartum home visitation from doulas, and support from doulas at the hospital during labor, delivery, and with early breastfeeding. Additionally, these participants receive longer-term home visiting services from family support workers during pregnancy and after the birth.
  Interventions: Behavioral: Doula Home Visiting
- Case Management (Active Comparator): Mothers in the comparison group receive low intensity case management services during pregnancy and following the birth.
  Interventions: Behavioral: Case management

INTERVENTIONS:
Behavioral: Doula Home Visiting — The intervention is a doula enhancement to evidence-based home visiting services. Doulas provide home visits during pregnancy and for the first six weeks postpartum, which focus on prenatal health, preparation for childbirth, bonding with the baby, and breastfeeding education. Family support workers provide longer term home visiting services. These home visits focus on sensitive and responsive parenting, early infant care, bonding with the baby, child health and development, and maternal mental health.
  Arms: Doula Home Visiting
Behavioral: Case management — Mothers are offered two prenatal and two postpartum case management meetings to assess whether mothers' basic needs (housing, nutrition, health care, mental health) are being met and make appropriate referrals.
  Arms: Case Management

SUMMARY:
The purpose of this randomized controlled trial is to examine whether evidence-based home visiting programs enhanced by doula services have effects on positive parenting practices, breastfeeding, and child and maternal health outcomes.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the impact of doula enhanced evidence-based home visiting programs for young mothers in Illinois. Mothers in the intervention group receive home visits from doulas during pregnancy and in the first few weeks postpartum, and doulas provide mothers with support at the hospital during labor, delivery, and with early breastfeeding. Additionally, mothers in the intervention group receive prenatal and long-term postpartum home visitation services through an evidence-based home visiting program, such as Parents as Teachers and Healthy Families Illinois. Mothers in the comparison group receive a less intensive case management service.

Four existing doula home visiting programs located in economically distressed communities in Illinois were selected for participation in the study. At each site, young pregnant women are recruited for participation in the study, provide informed consent, and complete a baseline interview in their homes during mid-pregnancy. At completion of the baseline interview, mothers are randomly assigned to either the doula home visiting intervention group or the case management comparison group.

At 37 weeks of pregnancy, and at 3 weeks-, 3 months-, 13 months-, and 30 months, and 4 years postpartum, mothers are interviewed in their homes on topics including pregnancy, parenting, health, mental health, feeding practices, employment/education, and relationships. Additionally, at all postpartum visits, mothers are videorecorded interacting with their infants. At the 13 month, 30 month, and 4 year followup sessions, children of the study participants are administered developmental and behavioral assessments.

Based on prior studies of doula services and the goals of doula enhanced home visiting programs, a variety of outcomes are assessed at followup time points. These outcomes include prenatal medical care, prenatal bonding with infant, feelings of efficacy during labor, anesthesia use during labor, breastfeeding, positive parenting behaviors, parenting attitudes and stress, infant health, maternal health, maternal depressive symptoms, and child behavior and development.

ELIGIBILITY:
Inclusion Criteria:

* pregnant and between 12 and 34 weeks gestation
* live within the catchment area of a program site
* between ages of 14-24
* English or Spanish speaking

Exclusion Criteria:

* ward of the Department of Children and Family Services (DCFS)
* under supervision of juvenile justice system
* planning to give up custody of infant
* pregnancy result of sexual assault

Ages: 14 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 312 (Actual)
Dates: Start 2011-11; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
National Institute of Child Health and Human Development (NICHD) mother-child interaction measures | 3 weeks postpartum
  Videotaped interactions between mothers and infants coded by masked observers for maternal sensitivity, intrusiveness, detachment, stimulation of cognitive development, positive and negative regard for the child, and flatness of affect.
Breastfeeding initiation | 3 weeks postpartum

SECONDARY OUTCOMES:
Breastfeeding duration | 3 week, 3 month, and 13 months postpartum
Maternal Antenatal Attachment Scale (MAAS) | 37 weeks of pregnancy
  The MAAS is a self-report scale that assesses a mother's emotional bond with her unborn infant.
Center for Epidemiologic Studies Depression Scale (CES-D) | 37 weeks pregnancy, and 3 weeks, 3 months, 13 months, 30 months, and 4 years postpartum
  The CES-D is a self report scale that measures symptoms of depression experienced in the past week.
Labour Agentry Scale | 3 weeks postpartum
  The Labour Agentry Scale is a self-report questionnaire that measures maternal feelings of efficacy during labor.
Use of labor analgesia | 3 weeks postpartum
Maternal Postnatal Attachment Scale (MPAS) | 3 weeks postpartum
  The MPAS is a self-report measure used to assess the quality of mother to infant attachment.
Parenting Stress Inventory (PSI) | 3 weeks, 3 months, 13 months, 30 months, and 4 years postpartum
  The PSI is a self report scale that assesses parenting stress and parent perceptions of the difficult of her child
Timing of solid food introduction | 3 weeks, 3 months, and 13 months postpartum
Knowledge of Infant Development Inventory (KIDI) | 3 months,13 months, and 30 months postpartum
  The KIDI is a self report questionnaire that assesses parent knowledge of parenting practices, infant behavior, and child development.
Infant/child ER visits | 3 weeks, 3 months, 13 months, 30 months, and 4 years postpartum
  Mother report of number of infant/child emergency room visits and reasons for visits
Infant/child immunizations | 13 months, 30 months, and 4 years postpartum
  Mother report of whether child is up to date on immunizations
Infant/child hospitalizations | 3 weeks, 3 months, 13 months, 30 months, and 4 years postpartum
  Mother report of number of infant/child hospitalizations and reasons for hospitalizations
Adult Adolescent Parenting Inventory (AAPI) | 3 months, 13 months, 30 months, and 4 years postpartum
  The AAPI is a self report scale that measures appropriate parenting attitudes.
Preschool Language Scales-5 (PLS-5) | 13 months postpartum
  The PLS-5 is an interactive assessment that measures children's auditory comprehension and expressive language. Trained assessors blind to intervention status administer the test to children of study participants.
Mullen Scales of Early Learning - Visual Reception | 13 months and 30 months postpartum
  The visual reception subscale of the Mullen measures children's ability to process information using patterns, sequencing, and memory. Trained assessors blind to intervention status administer the test to children of study participants.
Infant Toddler Social and Emotional Assessment (ITSEA) | 13 months and 30 months postpartum
  The ITSEA is a parent report scale that assesses problem behaviors and social competence of infants and toddlers.
Subsequent pregnancy | 3 month,13 months, 30 months, and 4 years postpartum
  Mothers report on whether they are currently pregnant
Parent-Child Conflict Tactics Scales (CTS PC) | 13 months, 30 months, and 4 years postpartum
  The CTS-PC is a parent report scale that measures how often parents use various forms of discipline and punishment with their children.
National Institute of Child Health and Human Development (NICHD) mother-child interaction measures. | 3 months, 13 months, and 30 months postpartum
  Videotaped interactions between mothers and infants coded by masked observers for maternal sensitivity, intrusiveness, detachment, stimulation of cognitive development, positive and negative regard for the child, and flatness of affect.
Woodcock-Johnson III Tests of Achievement | 4 years postpartum
  The WJ-III measures child achievement in reading readiness and quantitative skills

CONTACTS AND LOCATIONS:
Overall Officials: Sydney L Hans, PhD, Principal Investigator — The University of Chicago, School of Social Service Administration

REFERENCES:
- [Background] Hans SL, Edwards RC, Zhang Y. Randomized Controlled Trial of Doula-Home-Visiting Services: Impact on Maternal and Infant Health. Matern Child Health J. 2018 Oct;22(Suppl 1):105-113. doi: 10.1007/s10995-018-2537-7. PMID 29855838
- [Background] Hans SL, Edwards RC, Zhang Y. Correction to: Randomized Controlled Trial of Doula-Home-Visiting Services: Impact on Maternal and Infant Health. Matern Child Health J. 2018 Oct;22(Suppl 1):125. doi: 10.1007/s10995-018-2626-7. PMID 30128724
- [Background] Edwards RC, Vieyra Y, Hans SL. Maternal support for infant learning: Findings from a randomized controlled trial of doula home visiting services for young mothers. Early Childhood Research Quarterly. 2020; 51: 26-38.